CLINICAL TRIAL: NCT06854523
Title: Assessing Coronary Non-Culprit Plaque Early with Start of PCSK9 Inhibitors in Acute Myocardial Infarction
Brief Title: Assessing Coronary Non-Culprit Plaque Early with Start of PCSK9 Inhibitors in Acute Myocardial Infarction (ACCESS-AMI)
Acronym: ACCESS-AMI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yun Dai Chen (Other)
Responsible Party: Sponsor-Investigator, Yun Dai Chen, professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCVD2030-6
Record Dates: First submitted 2024-10-14; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-09

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Pericoronary artery fat attenuation index; Index of Plaque Attenuation; PCSK9 Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCSK9 inhibitor group (Experimental): In this group, patients will receive PCSK9 inhibitor treatment
  Interventions: Drug: PCSK9 inhibitor; Behavioral: Blood lipid levels meet the recommended guidelines
- Statin+ezetimibe group (Active Comparator): In this group, patients will receive statin and ezetimibe treatment
  Interventions: Drug: Statin+ezetimibe; Behavioral: Blood lipid levels don't meet the recommended guidelines

INTERVENTIONS:
Drug: PCSK9 inhibitor — The patient used Trastuzumab 150mg within 24 hours before or after PCI, and then every two weeks for 12 months
  Arms: PCSK9 inhibitor group
Drug: Statin+ezetimibe — The patient used statins and ezetimibe within 24 hours before or after PCI, and then once a day for 12 months
  Arms: Statin+ezetimibe group
Behavioral: Blood lipid levels meet the recommended guidelines — Early use of intensified lipid-lowering therapy during hospitalization led to a rapid decrease in blood lipids and met the recommended guidelines.
  Arms: PCSK9 inhibitor group
Behavioral: Blood lipid levels don't meet the recommended guidelines — The patient did not receive intensified lipid-lowering treatment during hospitalization or did not meet the recommended guidelines for blood lipids
  Arms: Statin+ezetimibe group

SUMMARY:
This study is planned to start on January 2024.

The goal of this clinical trial is to learn whether the perioperative administration (within 24 hours before or after primary PCI) of PCSK9 inhibitors can ameliorate plaque progression and adverse outcomes in patients with acute myocardial infarction (AMI). The main questions it aims to answer are:

Can perioperative PCSK9 inhibition improve the plaque stability and inflammation of perivascular adipose tissue (index of plaque attenuation（IPA ）and perivascular fat attenuation index（FAI）) of non-target lesions? Researchers will compare PCSK9 inhibitors with statin plus ezetimibe therapy to evaluate the potential of PCSK9 inhibitors in mitigating the progression of non-target lesion plaques and reducing adverse cardiovascular events in patients with AMI.

Participants will:

Take PCSK9 inhibitors every two weeks or daily statin plus ezetimibe therapy. Conduct a follow-up examination with optical coherence tomography (OCT) or coronary computed tomography angiography (CTA) after 12 months.

Record the occurrence of major adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Admitted to hospital for acute myocardial infarction (STEMI, NSTEMI) and successfully underwent PCI of the infarct vessel.
3. Coronary angiography revealed two non-infarct-related arteries with non-blocking lesions (diameter stenosis of 40-70%).
4. Able to sign informed consent.
5. Willing to undergo 1-year follow-up.

Exclusion Criteria:

1. Left main artery disease or severe coronary artery calcification;
2. Hemodynamic instability or uncontrolled arrhythmia;
3. History of coronary artery bypass;
4. severe renal insufficiency, active liver disease or liver insufficiency, hematological disease, metabolic or endocrine dysfunction, systemic infection, active malignant tumor and other potentially life-threatening diseases, or the expected survival time is < 1 year;
5. Received any PCSK9 inhibitor treatment within the previous 3 months;
6. Pregnant or nursing women or women planning pregnancy;
7. The researcher determined that it was not suitable for inclusion in the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Index of Plaque Attenuation (IPA) measured by OCT for non-culprit lesions at baseline and 12 months of follow-up. | 12 months
  IPA is a quantitative analysis tool based on OCT technology to evaluate plaque stability.
Changes in pericoronary artery fat attenuation index (FAI) measured by CCTA for non-culprit lesions at baseline and 12 months of follow-up | 12 months
  FAI is a quantitative indicator of inflammation in perivascular adipose tissue measured by CCTA.

SECONDARY OUTCOMES:
Progress of target lesion plaques | 12 months
  To assess plaque progression, OCT evaluation will include fiber cap thickness, lipid core amplitude, minimum lumen area, and minimum lumen diameter. CCTA evaluation will include CAD-RADS grade , plaque volume, plaque properties, calcification score, epicardial fat volume and plaque attenuation.
  Notes: CAD-RADS indicates Coronary Artery Disease-Reporting and Data System, which range from 0 to 5. The higher CAD-RADS grade, the more severe of the coronary stenosis.
The overall incidence of the first major adverse cardiovascular events (MACEs) within 12 months in different treatment groups | 12 months
  MACEs was defined as the composite of myocardial infarction, ischemic stroke, cardiovascular death and coronary revascularization
The proportion of LDLC at each visit node that meets the recommended guidelines and the changes compared to baseline | 1week；1months；3 months； 6 months; 9 months; 12 months
Changes in inflammatory factors (interleukin 6, C reaction protein) at each visit node compared to baseline | 1week；1months；3 months； 6 months; 9 months; 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital [, Beijing